CLINICAL TRIAL: NCT04309370
Title: Interactions of Fronto-Parietal High Frequency Repetitive Transcranial Magnetic Stimulation on Anterior Cingulate Cortex Activation in Schizophrenia
Brief Title: Interactions of Fronto-Parietal High Frequency rTMS on Anterior Cingulate Cortex Activation in Schizophrenia
Acronym: rTMS-FPCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Tom Hummer, Associate Research Professor of Psychiatry, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1909015657
Record Dates: First submitted 2019-12-20; First posted 2020-03-16 (Actual); Results first posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Schizophrenia
Keywords: schizophrenia; psychosis; early phase psychosis; rTMS
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 20 Hz rTMS targeting the LDLPFC first, then 20 Hz rTMS targeting the LSPC (Experimental)
  Interventions: Device: 20 Hz rTMS
- 20 Hz rTMS Targeting the LSPC first, then 20 Hz rTMS Targeting the LDLPFC (Experimental)
  Interventions: Device: 20 Hz rTMS

INTERVENTIONS:
Device: 20 Hz rTMS — Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive neuromodulation technique that received FDA clearance for use in treatment resistant major depressive disorder in 2008. rTMS utilizes the application of a repetitively pulsed magnetic field over the scalp to induce an electric field within a discrete area of the cerebral cortex. This electric field results in altered ion flow across the neuronal cellular membrane and ultimately changes in neuronal polarization. rTMS modulates cortical activation depending on the stimulation parameters used. Physiological studies have provided evidence that suggests that high-frequency (HF) rTMS produces an increase in local cortical excitability. Studies have also demonstrated that rTMS may increase or decrease functional connectivity between separate but related cortical structures, utilizing high and low frequency stimulation, respectively.

SUMMARY:
This will be a single site pilot study. 20 subjects with EPP (Early Phase Psychosis), defined as medical record documentation of the onset of clinically significant psychotic symptoms within the past 10 years, will be enrolled. Prior to randomization subjects will undergo fMRI (Functional Magnetic Resonance Imaging) during CC (Cognitive Control) task (Stroop Color-Word paradigm) and resting-state paradigms. This baseline scan will also include a high-resolution structural sequence for neuronavigation purposes. Then, on two separate days, each occurring one-week apart, subjects will receive one session of excitatory (20 Hz) (Hertz) rTMS (Repetitive Transcranial Magnetic Stimulation) targeting the LDLPFC (Left Dorsolateral Prefrontal Cortex) and one session targeting the LSPC (Left Superior Parietal Cortex). The order of stimulation sites will be randomized and counter-balanced. Immediately following each session, subjects will undergo repeat fMRI during CC and RS (Resting State) paradigms. Investigators will also examine the effect of rTMS on CC performance.

DETAILED DESCRIPTION:
In spite of existing work studying rTMS as a treatment modality in schizophrenia, there are no studies that have examined the effects of rTMS targeting superficial CCN (Cognitive Control Network) structures (LDLPFC and LSPC) on ACC (Anterior Cingulate Cortex) activity or CCN connectivity in schizophrenia. It is also important to note that the vast majority of studies using rTMS in schizophrenia have examined chronic populations where confounds associated with prolonged duration of illness may be present. EPP is a desirable population to study because these individuals tend to have fewer psychiatric and physical comorbidities and less antipsychotic drug exposure, all of which are factors that may confound investigations of new treatment interventions for this illness. In light of the significant unmet medical need associated with schizophrenia and the grave clinical effect of disrupted CC in the illness, rTMS modulating the ACC, and potentially CCN circuitry, represents an unexplored and novel potential treatment option.

The goal of this project is to utilize HF (20 Hz) rTMS, in conjunction with functional magnetic resonance imaging (fMRI), to provide evidence that rTMS targeting superficial CCN structures (LDLPFC and LSPC) modulates: 1) activation in the ACC during in-scanner CC task performance and 2) functional connectivity between the CCN structures during in-scanner CC task performance. This study will provide vital preliminary data on target engagement informing future clinical trials seeking to investigate rTMS as a novel treatment for CC impairment in schizophrenia. This study will also seek to refine the understanding of the brain circuitry that mediates the potential pro-CC effects of rTMS through the use of fMRI at baseline and following the course of rTMS administration.

ELIGIBILITY:
Inclusion Criteria:

1. Between 18 and 40 years of age
2. Within 10 years of illness onset as defined by entry into treatment for psychotic symptoms
3. Able to give informed consent
4. Willing and able to adhere to the study schedule
5. Mini-International Neuropsychiatric interview (MINI)37-40 diagnosis of schizophrenia
6. Clinical stability defined by:

   1. Subjects must not have experienced an exacerbation of their illness within 4 weeks prior to randomization, leading to an intensification of psychiatric care in the opinion of the investigator. Examples of intensification of care include, but are not limited to: inpatient hospitalization, day/partial hospitalization, outpatient crisis management, or psychiatric treatment in an emergency room AND
   2. Antipsychotic treatment stability for at least 4 weeks prior to randomization (no change in antipsychotic dosing or addition of new antipsychotic medication)

Exclusion Criteria:

1. Lifetime history of a seizure, excluding febrile seizures and those induced by substance withdrawal
2. First degree relative with idiopathic epilepsy or other seizure disorder
3. History of significant neurological illness
4. History of head trauma as defined by a loss of consciousness or a post-concussive syndrome
5. Pregnant or breast feeding
6. Known IQ < 70 based on subject report
7. Current acute, serious, or unstable medical conditions
8. Metallic objects planted in or near the head, including implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator, TENS unit, ventriculoperitoneal shunt, or cochlear implants
9. Contraindications to MRI or otherwise unable to tolerate MRI procedures
10. History of electroconvulsive therapy
11. Subjects taking clozapine
12. Subjects who have participated in a clinical trial with any pharmacological treatment intervention for which they received study-related medication in the 4 weeks prior to randomization
13. Subjects considered a high risk for suicidal acts - active suicidal ideation as determined by clinical interview OR any suicide attempt in 90 days prior to screening
14. Current DSM-5 diagnosis of alcohol or drug use disorder (excluding nicotine or caffeine)
15. Subjects who require concomitant treatment with prohibited medication, as specified in Attachment 2

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Hummer, PhD, Principal Investigator — Indiana University
Locations (2):
- United States (2):
  - IU Center for Neuroimaging, Indianapolis, Indiana
  - Prevention and Recovery Center for Early Psychosis, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 20 Hz rTMS Targeting the LDLPFC First, Then 20 Hz rTMS Targeting the LSPC | 20 Hz rTMS Targeting the LSPC First, Then 20 Hz rTMS Targeting the LDLPFC
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 20 Hz rTMS Targeting the LDLPFC First, Then 20 Hz rTMS Targeting the LSPC | 20 Hz rTMS Targeting the LSPC First, Then 20 Hz rTMS Targeting the LDLPFC | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.9 (2.1) | 27.2 (5.1) | 26.5 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 7 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in BOLD Signal in Anterior Cingulate Cortex
Description: Effects of rTMS on anterior cingulate cortex functional activation as measured by blood oxygen level dependent (BOLD) signal change scores during cognitive control Mismatch trials vs. Match trials (i.e., Mismatch - Match). The BOLD signal is measured during a functional magnetic resonance imaging (fMRI) scan and reflects the level of brain activity in the region. Change is calculated as difference between the Mismatch-Match signal at baseline and 30-60 minutes following the intervention. Higher scores indicate a larger increase in brain activity following the intervention.
Time Frame: 1 day
Measure: Mean (95% Confidence Interval); unit: BOLD signal change (Mismatch vs. Match)
Groups:
- 20 Hz rTMS Targeting the Left DLPFC: Subjects will receive a 20 Hz repetitive transcranial magnetic stimulation (rTMS) directed at the left dorsolateral prefrontal cortex (DLPFC) at 110% of motor threshold, with 60 trains, 20 pulses per train, with 1200 pulses over 21 minutes.
- 20 Hz rTMS Targeting the Left Superior Parietal Cortex: Subjects will receive a 20 Hz repetitive transcranial magnetic stimulation (rTMS) directed at the left superior parietal cortex at 110% of motor threshold, with 60 trains, 20 pulses per train, with 1200 pulses over 21 minutes.
Arm/Group | 20 Hz rTMS Targeting the Left DLPFC | 20 Hz rTMS Targeting the Left Superior Parietal Cortex
Number analyzed (Participants) | 14 | 14
BOLD signal change (Mismatch vs. Match) | -0.0188 [-0.176 to 0.187] | 0.0124 [-0.086 to 0.152]

2. Primary Outcome: Change in Cognitive Control Network Functional Connectivity
Description: The outcome reflects changes in blood oxygen level dependent (BOLD) functional connectivity with anterior cingulate cortex (ACC) and the left dorsolateral prefrontal cortex (LDLPFC) and left superior parietal cortex (LSPC). Functional connectivity is calculated as the Fisher's transformation of the correlation coefficient of the BOLD time series in the ACC with the time series in each target region. Therefore, functional connectivity reflects how similar brain activity is between the target regions (LDLPFC and LSPC) and the ACC, with higher scores indicating greater connectivity. Outcome scores are changes in this connectivity between baseline and 30-60 minutes following the rTMS intervention targeting LDLPFC or LSPC. Positive scores indicate stronger connectivity following rTMS in the cognitive control network.
Time Frame: 1 day
Measure: Mean (95% Confidence Interval); unit: Change in correlation
Arm/Group | 20 Hz rTMS Targeting the Left DLPFC | 20 Hz rTMS Targeting the Left Superior Parietal Cortex
Number analyzed (Participants) | 14 | 14
Change in correlation | -0.006 [-0.348 to 0.286] | -0.01 [-0.262 to 0.121]

ADVERSE EVENTS:
Time Frame: 1 month
Description: Investigator evaluated for adverse events at every visit
Groups:
- 20 Hz rTMS Targeting the LDLPFC; 20 Hz rTMS Targeting the LSPC: 20 Hz rTMS: Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive neuromodulation technique that received FDA clearance for use in treatment resistant major depressive disorder in 2008. rTMS utilizes the application of a repetitively pulsed magnetic field over the scalp to induce an electric field within a discrete area of the cerebral cortex. This electric field results in altered ion flow across the neuronal cellular membrane and ultimately changes in neuronal polarization. rTMS modulates cortical activation depending on the stimulation parameters used. Physiological studies have provided evidence that suggests that high-frequency (HF) rTMS produces an increase in local cortical excitability. Studies have also demonstrated that rTMS may increase or decrease functional connectivity between separate but related cortical structures, utilizing high and low frequency stimulation, respectively.
Arm/Group | 20 Hz rTMS Targeting the LDLPFC | 20 Hz rTMS Targeting the LSPC
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 2/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20 Hz rTMS Targeting the LDLPFC (N=14) | 20 Hz rTMS Targeting the LSPC (N=14)
Application site discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT04309370/Prot_SAP_000.pdf